CLINICAL TRIAL: NCT02287376
Title: A Phase 4, Open-Label Study of the Pharmacokinetics and Safety of Cambia® (Diclofenac Potassium for Oral Solution) for the Acute Treatment of Migraine Attacks With or Without Aura in Pediatric Subjects (Ages 12-17 Years)
Brief Title: Pharmacokinetics & Safety of Cambia® in Migraine With or Without Aura in 12-17 Year Olds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81-0076
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Migraine
Keywords: Migraine with and without aura
MeSH Terms: conditions — Migraine Disorders | interventions — Diclofenac; Solutions

ARMS (1):
- Diclofenac Potassium (Experimental): Diclofenac Potassium for Oral Solution 50 mg
  Interventions: Drug: Diclofenac Potassium for Oral Solution

INTERVENTIONS:
Drug: Diclofenac Potassium for Oral Solution — NSAID
  Other Names: Cambia

SUMMARY:
Study Objectives:

1. The primary objective is to characterize the pharmacokinetics of a single oral administration of 50 mg Cambia in pediatric subjects, ages 12-17 years with a diagnosis of episodic migraine with or without aura.
2. The secondary objectives are to determine:

   1. The safety and tolerability of Cambia from a single dose
   2. Three-month safety evaluation of Cambia in outpatient usage in this population

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥12 and ≤17 years of age at screening.
2. Subject diagnosed with episodic migraine with or without aura for at least 3 months (migraine defined based on the International classification of headache disorders-II 1.2.1 or 1.1).
3. Subject has 14 or fewer headache days per month.
4. Subject receiving prophylactic treatment for migraine may be included.
5. If female, is not of childbearing potential (defined as premenarchal) or if of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Study Day 1, if the Screening visit and Day 1 are not on the same day, and must use medically acceptable methods of birth control as listed below and agrees to continue its use throughout the study:1) hormonal methods (e.g., oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full menstrual cycle before study drug administration), 2) Total abstinence from sexual intercourse since the last menses before study drug administration, 3) intrauterine device, 4) double-barrier method (e.g., condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream).
6. Subject's legally authorized representative (e.g., parent, guardian) must voluntarily sign and date an informed consent form (ICF) that is approved by an Institutional Review Board (IRB), and the subject must sign an assent (if appropriate), before the commencement of any study assessment.
7. Subject's legally authorized representative (e.g., parent, guardian) and subject (if appropriate), is able to read and understand the study procedures and requirements and adhere to the protocol requirements and procedures.

Exclusion Criteria:

1. Subject has a known history of allergic reaction, hypersensitivity, or clinically significant intolerance to diclofenac, aspirin, or any nonsteroidal anti inflammatory drugs (NSAIDs); history of NSAID induced bronchospasm (subjects with the triad of asthma, nasal polyps, and chronic rhinitis are at greater risk for bronchospasm and should be considered carefully); or hypersensitivity, allergy, or significant reaction to the non-active ingredients of the study medication.
2. Subject is pregnant or lactating or considered at risk of pregnancy.
3. Subject has been under an inconsistent dosing regimen of prophylactic treatment for migraine.
4. Subject has headache symptoms likely due to, or aggravated by, traumatic injury to the head or neck region, such as whiplash, within the last six months;
5. Subject has or is suspected of having a secondary headache.
6. Subject has significant abnormal findings during the neurological exam at screening.
7. Subject has a history of any GI event (e.g., perforation, obstruction, bleed) before Screening that, in the opinion of the investigator, would make the subject unsuitable for study participation.
8. Subject is receiving any medication that, in the opinion of the investigator, may cause a clinically significant condition when used concomitantly with diclofenac (e.g., aspirin, anticoagulants, ACE inhibitors, methotrexate, cyclosporine, furosemide, lithium).
9. Subject is and has been receiving a medication that is known to strongly inhibit and/or induce cytochrome P450 2C9 such that it might unpredictably affect the pharmacokinetics of diclofenac (e.g., fluconazole, amiodarone, oxandrolone, sulfipyrazone as inhibitors and rifampin as an inducer).
10. Subject has any condition or any laboratory abnormality that would, in the opinion of the investigator, contraindicate study participation.
11. Subject has impaired liver function (e.g., alanine aminotransferase [ALT] ≥ 3 times the upper limit of normal [ULN] or bilirubin ≥ 3 times ULN), known active hepatic disease (e.g., hepatitis), or evidence of clinically significant liver disease or other condition affecting the liver that may suggest the potential for an increased susceptibility to hepatic toxicity with oral diclofenac exposure.
12. Subject has any history of renal disease that, in the opinion of the investigator, would contraindicate study participation; or subject has significantly impaired renal function as evidenced by an estimated GFR of ≤60 ml/min/1.73m2.
13. Subject is considered by the investigator, for any reason (including, but not limited to the risks described as precautions, warnings, and contraindications in the Prescribing Information for Cambia), to be an unsuitable candidate to receive the study medication.
14. Subject has a history of laboratory test results obtained within 6 months before the Screening visit that show the presence of HIV, hepatitis B surface antigen, hepatitis C antibody, or active hepatitis A immunoglobulin M.
15. Subject is currently receiving any medication that is contraindicated for use concomitantly with diclofenac (refer to the products' professional labeling) or the subject has not undergone a washout period of at least 5-6 half-lives of PK or PD, whichever is longer, for these medications.
16. Subject has a known or suspected history of alcohol use and or drug/ substance abuse or misuse within 2 years before Screening; or evidence of tolerance or physical dependence before study medication administration.
17. Subject has a documented history of a medical condition that, in the opinion of the investigator, would compromise the subject's ability to absorb, metabolize, or excrete diclofenac, including (but not limited to) intractable nausea and/or vomiting and/or severe GI narrowing (pathologic or iatrogenic).
18. Subject has received any investigational product or device within 30 days before the Screening, or is scheduled to receive an investigational device or another investigational drug (other than Cambia) during the course of this study.
19. Subject is a relative of a member of the study site staff or Sponsor directly involved in this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tampa, Florida
  - Amherst, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Cambia®: Diclofenac Potassium for Oral Solution (NSAID), 50 mg
Period: Overall Study
Arm/Group | Cambia®
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Outcome (1 of 6)
Description: • Cmax: maximum concentration (ng/mL)
Time Frame: 6 hours (pre-dose, 5, 10, 15, 20, 30, 40, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: The PK population included all subjects in the Safety population who have at least 1 time point with quantifiable study drug concentration after dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cambia®
Number analyzed (Participants) | 25
ng/mL
  Cmax (ng/mL) | 1411.96 (846.208)
  pre-dose concentrations (ng/mL) | 0.00 (0.000)
  5 min post-dose concentrations (ng/mL) | 649.78 (1008.783)
  10 min post-dose concentrations (ng/mL) | 1123.88 (881.619)
  15 min post-dose concentrations (ng/mL) | 1247.72 (824.194)
  20 min post-dose concentrations (ng/mL) | 1084.52 (575.825)
  30 min post-dose concentrations (ng/mL) | 855.92 (469.835)
  40 min post-dose concentrations (ng/mL) | 629.96 (295.361)
  60 min post-dose concentrations (ng/mL) | 535.44 (295.222)
  2 hrs post-dose concentrations (ng/mL) | 164.25 (107.706)
  4 hrs post-dose concentrations (ng/mL): number analyzed (Participants) | 24
  4 hrs post-dose concentrations (ng/mL) | 40.20 (25.285)
  6 hrs post-dose concentrations (ng/mL): number analyzed (Participants) | 24
  6 hrs post-dose concentrations (ng/mL) | 14.26 (7.507)

2. Primary Outcome: Pharmacokinetics Outcome (2 of 6)
Description: • tmax: time to maximum concentration (min)
Time Frame: 6 hours (pre-dose, 5, 10, 15, 20, 30, 40, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Cambia®
Number analyzed (Participants) | 25
min | 18.00 (11.551)

3. Primary Outcome: Pharmacokinetics Outcome (3 of 6)
Description: • λz: elimination rate constant associated with the terminal (log linear) portion of the curve (1/min)
Time Frame: 6 hours (pre-dose, 5, 10, 15, 20, 30, 40, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/min
Arm/Group | Cambia®
Number analyzed (Participants) | 24
1/min | 0.01 (0.002)

4. Primary Outcome: Pharmacokinetics Outcome (4 of 6)
Description: • t1/2: terminal elimination half-life (min)
Time Frame: 6 hours (pre-dose, 5, 10, 15, 20, 30, 40, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Cambia®
Number analyzed (Participants) | 24
min | 66.79 (9.193)

5. Primary Outcome: Pharmacokinetics Outcome (5 of 6)
Description: • AUC 0-t: area under the concentration-time curve from time 0 to last time point (t) where diclofenac could be measured (min*ng/mL)
Time Frame: 6 hours (pre-dose, 5, 10, 15, 20, 30, 40, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Cambia®
Number analyzed (Participants) | 25
min*ng/mL | 82920.03 (25327.634)

6. Primary Outcome: Pharmacokinetics Outcome (6 of 6)
Description: • AUC 0-∞: area under the concentration-time curve from time 0 to infinity (∞) (min*ng/mL)
Time Frame: 6 hours (pre-dose, 5, 10, 15, 20, 30, 40, and 60 min, and 2, 4, and 6 hrs post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Cambia®
Number analyzed (Participants) | 24
min*ng/mL | 84388.75 (25993.623)

7. Secondary Outcome: Safety Outcome (1 of 7)
Description: • Treatment emergent AEs (TEAEs)
Time Frame: 3 months (time of first dose of study medication taken to 30 days after the last dose of study medication taken)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Participants | 10

8. Secondary Outcome: Safety Outcome (2 of 7)
Description: • Serious adverse events (SAEs)
Time Frame: 3 months (signed informed consent/assent to 30 days post Day 90 or last dose of study medication taken)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Participants | 1

9. Secondary Outcome: Safety Outcome (3 of 7)
Description: • Withdrawals due to AEs
Time Frame: 3 months (signed informed consent/assent to 30 days after the last dose of study medication taken)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Participants | 0

10. Secondary Outcome: Safety Outcome (4 of 7)
Description: • Deaths
Time Frame: 3 months (signed informed consent/assent to 30 days post Day 90 or last dose of study medication taken)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Participants | 0

11. Secondary Outcome: Safety Outcome (5.1 of 7)
Description: • Changes in vital sign measurements: Temperature (degrees C).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
  The data presented are changes from baseline to the final visit. Baseline is defined as the last measurement taken before first treatment with study drug.
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Cambia®
Number analyzed (Participants) | 25
degrees C
  Baseline (degrees C) | 36.52 (0.569)
  Final Visit (degrees C) | 36.72 (0.499)
  Change from Baseline to Final Visit (degrees C) | 0.20 (0.491)

12. Secondary Outcome: Safety Outcome (5.2 of 7)
Description: • Changes in vital sign measurements: Heart Rate (beats/min).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Cambia®
Number analyzed (Participants) | 25
beats/min
  Baseline (beats/min) | 74.6 (12.41)
  Final Visit (beats/min) | 74.7 (9.23)
  Change from Baseline to Final Visit (beats/min) | 0.2 (10.95)

13. Secondary Outcome: Safety Outcome (5.3 of 7)
Description: • Changes in vital sign measurements: Respiratory Rate (breaths/min).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Cambia®
Number analyzed (Participants) | 25
breaths/min
  Baseline (breaths/min) | 15.4 (1.23)
  Final Visit (breaths/min) | 15.6 (0.82)
  Change from Baseline to Final Visit (breaths/min) | 0.1 (1.42)

14. Secondary Outcome: Safety Outcome (5.4 of 7)
Description: • Changes in vital sign measurements: Systolic Blood Pressure (mmHg).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mm Hg
  Baseline (mm Hg) | 112.7 (11.71)
  Final Visit (mm Hg) | 109.6 (9.83)
  Change from Baseline to Final Visit (mm Hg) | -3.1 (14.27)

15. Secondary Outcome: Safety Outcome (5.5 of 7)
Description: • Changes in vital sign measurements: Diastolic Blood Pressure (mmHg).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mm Hg
  Baseline (mm Hg) | 68.8 (8.78)
  Final Visit (mm Hg) | 67.1 (7.07)
  Change from Baseline to Final Visit (mm Hg) | -1.7 (9.62)

16. Secondary Outcome: Safety Outcome (6.1 of 7)
Description: • Changes in clinical laboratory results: Hematology - Hematocrit (L/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
L/L
  Baseline (L/L) | 0.388 (0.0329)
  Final Visit (L/L) | 0.408 (0.0344)
  Change from Baseline to Final Visit (L/L) | 0.020 (0.0190)

17. Secondary Outcome: Safety Outcome (6.2 of 7)
Description: • Changes in clinical laboratory results: Hematology - Hemoglobin (g/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
g/L
  Baseline (g/L) | 128.000 (11.4419)
  Final Visit (g/L) | 132.720 (11.6638)
  Change from Baseline to Final Visit (g/L) | 4.720 (5.4430)

18. Secondary Outcome: Safety Outcome (6.3 of 7)
Description: • Changes in clinical laboratory results: Hematology - Platelet Count (Cells * 10^9/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Cells * 10^9/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Cells * 10^9/L
  Baseline (Cells * 10^9/L) | 233.640 (43.4855)
  Final Visit (Cells * 10^9/L) | 244.960 (47.0049)
  Change from Baseline to Final Visit (Cells*10^9/L) | 11.320 (42.3642)

19. Secondary Outcome: Safety Outcome (6.4 of 7)
Description: • Changes in clinical laboratory results: Hematology - White Blood Cells (Cells * 10^9/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Cells * 10^9/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Cells * 10^9/L
  Baseline (Cells * 10^9/L) | 6.512 (1.9935)
  Final Visit (Cells * 10^9/L) | 6.262 (1.4957)
  Change from Baseline to Final Visit (Cells*10^9/L) | -0.249 (2.0634)

20. Secondary Outcome: Safety Outcome (6.5 of 7)
Description: • Changes in clinical laboratory results: Hematology - Basophils (%).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % Basophils
Arm/Group | Cambia®
Number analyzed (Participants) | 25
% Basophils
  Baseline (% Basophils) | 0.324 (0.3829)
  Final Visit (% Basophils) | 0.350 (0.3766)
  Change from Baseline to Final Visit (% Basophils) | 0.026 (0.5190)

21. Secondary Outcome: Safety Outcome (6.6 of 7)
Description: • Changes in clinical laboratory results: Hematology - Eosinophils (%).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % Eosinophils
Arm/Group | Cambia®
Number analyzed (Participants) | 25
% Eosinophils
  Baseline (% Eosinophils) | 2.730 (2.0728)
  Final Visit (% Eosinophils) | 2.036 (1.6519)
  Change from Baseline to Final Visit(% Eosinophils) | -0.694 (1.7186)

22. Secondary Outcome: Safety Outcome (6.7 of 7)
Description: • Changes in clinical laboratory results: Hematology - Neutrophils (%).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % Neutrophils
Arm/Group | Cambia®
Number analyzed (Participants) | 25
% Neutrophils
  Baseline (% Neutrophils) | 54.530 (9.7221)
  Final Visit (% Neutrophils) | 57.932 (8.4095)
  Change from Baseline to Final Visit(% Neutrophils) | 3.402 (10.1083)

23. Secondary Outcome: Safety Outcome (6.8 of 7)
Description: • Changes in clinical laboratory results: Hematology - Lymphocytes (%).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % Lymphocytes
Arm/Group | Cambia®
Number analyzed (Participants) | 25
% Lymphocytes
  Baseline (% Lymphocytes) | 36.260 (8.9981)
  Final Visit (% Lymphocytes) | 33.745 (7.5260)
  Change from Baseline to Final Visit(% Lymphocytes) | -2.515 (9.1165)

24. Secondary Outcome: Safety Outcome (6.9 of 7)
Description: • Changes in clinical laboratory results: Hematology - Monocytes (%).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % Monocytes
Arm/Group | Cambia®
Number analyzed (Participants) | 25
% Monocytes
  Baseline (% Monocytes) | 6.030 (1.8765)
  Final Visit (% Monocytes) | 5.847 (1.7170)
  Change from Baseline to Final Visit (% Monocytes) | -0.183 (1.7852)

25. Secondary Outcome: Safety Outcome (6.10 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Albumin (g/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
g/L
  Baseline (g/L) | 43.800 (4.0415)
  Final Visit (g/L) | 47.200 (4.4441)
  Change from Baseline to Final Visit (g/L) | 3.400 (3.0277)

26. Secondary Outcome: Safety Outcome (6.11 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Alkaline Phosphatase (U/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
U/L
  Baseline (U/L) | 98.960 (85.0022)
  Final Visit (U/L) | 103.760 (89.5378)
  Change from Baseline to Final Visit (U/L) | 4.800 (11.4054)

27. Secondary Outcome: Safety Outcome (6.12 of 7)
Description: • Changes in clinical laboratory results: Chemistry - ALT (SGPT) (U/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
U/L
  Baseline (U/L) | 12.680 (5.7134)
  Final Visit (U/L) | 13.080 (5.1553)
  Change from Baseline to Final Visit (U/L) | 0.400 (2.0817)

28. Secondary Outcome: Safety Outcome (6.13 of 7)
Description: • Changes in clinical laboratory results: Chemistry - AST (SGOT) (U/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
U/L
  Baseline (U/L) | 17.240 (4.5760)
  Final Visit (U/L) | 18.040 (4.6947)
  Change from Baseline to Final Visit (U/L) | 0.800 (2.6615)

29. Secondary Outcome: Safety Outcome (6.14 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Bicarbonate (CO2) (mmol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mmol/L
  Baseline (mmol/L) | 23.400 (1.8028)
  Final Visit (mmol/L) | 23.920 (2.1970)
  Change from Baseline to Final Visit (mmol/L) | 0.520 (2.7099)

30. Secondary Outcome: Safety Outcome (6.15 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Bilirubin Total (umol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
umol/L
  Baseline (umol/L) | 9.029 (4.1454)
  Final Visit (umol/L) | 10.192 (5.5311)
  Change from Baseline to Final Visit (umol/L) | 1.163 (3.9107)

31. Secondary Outcome: Safety Outcome (6.16 of 7)
Description: • Changes in clinical laboratory results: Chemistry - BUN (Urea) (mmol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mmol/L
  Baseline (mmol/L) | 4.512 (1.0858)
  Final Visit (mmol/L) | 4.594 (1.2965)
  Change from Baseline to Final Visit (mmol/L) | 0.081 (1.0515)

32. Secondary Outcome: Safety Outcome (6.17 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Chloride (mmol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mmol/L
  Baseline (mmol/L) | 105.480 (1.9604)
  Final Visit (mmol/L) | 104.880 (2.7435)
  Change from Baseline to Final Visit (mmol/L) | -0.600 (2.1602)

33. Secondary Outcome: Safety Outcome (6.18 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Creatinine (umol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
umol/L
  Baseline (umol/L) | 66.760 (11.2603)
  Final Visit (umol/L) | 67.467 (10.7228)
  Change from Baseline to Final Visit (umol/L) | 0.707 (8.1866)

34. Secondary Outcome: Safety Outcome (6.19 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Glucose (mmol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mmol/L
  Baseline (mmol/L) | 4.758 (0.6037)
  Final Visit (mmol/L) | 4.483 (0.8590)
  Change from Baseline to Final Visit (mmol/L) | -0.275 (0.9215)

35. Secondary Outcome: Safety Outcome (6.20 of 7)
Description: • Changes in clinical laboratory results: Chemistry - LDH (U/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
U/L
  Baseline (U/L): number analyzed (Participants) | 17
  Baseline (U/L) | 157.882 (59.0824)
  Final Visit (U/L): number analyzed (Participants) | 24
  Final Visit (U/L) | 159.708 (41.5425)
  Change from Baseline to Final Visit (U/L): number analyzed (Participants) | 17
  Change from Baseline to Final Visit (U/L) | -0.882 (74.6064)

36. Secondary Outcome: Safety Outcome (6.21 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Potassium (mmol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mmol/L
  Baseline (mmol/L) | 3.964 (0.2215)
  Final Visit (mmol/L) | 4.060 (0.2784)
  Change from Baseline to Final Visit (mmol/L) | 0.096 (0.3007)

37. Secondary Outcome: Safety Outcome (6.22 of 7)
Description: • Changes in clinical laboratory results: Chemistry - Sodium (mmol/L).
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cambia®
Number analyzed (Participants) | 25
mmol/L
  Baseline (mmol/L) | 138.640 (1.0360)
  Final Visit (mmol/L) | 138.840 (1.5188)
  Change from Baseline to Final Visit (mmol/L) | 0.200 (1.6833)

38. Secondary Outcome: Safety Outcome (6.23 of 7)
Description: • Changes in clinical laboratory results: Urinalysis - pH.
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cambia®
Number analyzed (Participants) | 25
pH
  Baseline (pH) | 6.220 (0.7511)
  Final Visit (pH) | 6.300 (0.7773)
  Change from Baseline to Final Visit (pH) | 0.080 (0.8977)

39. Secondary Outcome: Safety Outcome (6.24 of 7)
Description: • Changes in clinical laboratory results: Urinalysis - Specific Gravity.
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Specific Gravity
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Specific Gravity
  Baseline (Specific Gravity) | 1.020 (0.0085)
  Final Visit (Specific Gravity) | 1.022 (0.0060)
  Change from Baseline to Final Visit (Spec.Gravity) | 0.002 (0.0081)

40. Secondary Outcome: Safety Outcome (7 of 7)
Description: • Physical examination findings including abnormal clinically significant findings
Time Frame: 3 months (signed informed consent/assent to the final visit)
Population: The Safety population included all subjects who have received at least 1 dose of study drug.
  The data presented is a clinically significant change from baseline to the final visit. Baseline is defined as the last measurement taken before first treatment with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cambia®
Number analyzed (Participants) | 25
Participants | 1

ADVERSE EVENTS:
Time Frame: 3 months (signed informed consent/assent to 30 days post Day 90 or last dose of study medication taken)
Description: The Safety population included all subjects who have received at least 1 dose of study drug.
Arm/Group | Cambia®
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cambia® (N=25)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Migraine (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cambia® (N=25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Motion Sickness (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and / or proprietary other than study data.